CLINICAL TRIAL: NCT04419012
Title: Polish Atrial Fibrillation (POL-AF) Registry
Acronym: POL-AF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jan Kochanowski University (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Iwona Gorczyca, MD, PhD, Principal Investigator, Jan Kochanowski University
Other Study IDs: 104/018
Record Dates: First submitted 2020-05-13; First posted 2020-06-05 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; anticoagulant treatment; apixaban; dabigatran; rivaroxaban; vitamin K antagonist; stroke prevention
MeSH Terms: conditions — Atrial Fibrillation | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with AF treated with VKA
  Interventions: Other: observation
- Patients with AF treated with NOAC
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
Evaluation of clinical characteristics and pharmacotherapy of hospitalized Polish patients with atrial fibrillation (AF).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common arrhythmia associated with increased cardiovascular mortality. An important element of management of patients with AF is anticoagulation to prevent thromboembolic events. Non-vitamin K oral anticoagulants (NOACs) and vitamin K antagonists (VKAs) are two main drugs groups used in thromboembolic events prevention.

Primary objective of the study is to assess the frequency of VKAs vs NOACs prescription in AF patients treatment of with OACs.

Secondary objective of the study are as follows: assessment of the frequency of appropriate/inappropriate OACs prescription in AF patients and assesment of the number of patients with AF treated with apixaban, dabigatran and rivaroxaban with high thromboembolism risk according to CHA2DS2-VASc score.

The POL-AF Registry is a multicenter prospective analysis of hospital records of patients with AF managed in ten cardiology centers.

Collected data will include demographics, type of AF (valvular and non-valvular, as well as paroxysmal, persistent and permanent), medical history, laboratory tests, echocardiographic parameters and concomitant medications.

Each patient will be evaluated regarding to common scales assessing risk of thromboembolic (CHA2DS2-VASc) and bleeding (HAS-BLED, modifiable and non-modifiable risk factors for bleeding in anticoagulated patients basing on the current guidelines for AF treatment) events.

ELIGIBILITY:
Inclusion Criteria:

- patients with AF hospitalized in a participating center during study period

Exclusion Criteria:

* hospitalisation for atrial fibrillation ablation
* death during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with AF hospitalized in a participating center during study period.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-01-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the frequency of VKAs vs NOACs prescription in AF patients treatment of with OACs. | Through the study completion, an average of 2 months.
  Compared data will include: frequency of VKAs vs NOACs prescriptions.

SECONDARY OUTCOMES:
Assessment of the frequency of appropriate/inappropriate OACs prescription in AF patients. | Through the study completion, an average of 2 months.
  Compared data will include: demographics, type of AF, medical history, baseline characteristics and concomitant medications.
Number of patients with AF treated with apixaban, dabigatran and rivaroxaban with high thromboembolism risk according to CHA2DS2-VASc (heart failure, hypertension, age, diabetes mellitus, stroke/TIA/thromboembolism, vascular disease and sex) score. | Through the study completion, an average of 2 months.
  The CHA2DS2-VAS score includes the following factors: heart failure, hypertension, age, diabetes mellitus, stroke/TIA/thromboembolism, vascular disease and sex.
  According to the CHA2DS2-VAS score, high thromboembolic risk means 2 points in men, 3 points in women.
  Data on the components of CHA2DS2-VASC are obtained from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Gorczyca, Md,PhD, Principal Investigator — Collegium Medicum, Jan Kochanowski University
Locations (1):
- Iwona Gorczyca, Kielce, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Uzieblo-Zyczkowska B, Krzesinski P, Maciorowska M, Gorczyca I, Jelonek O, Wojcik M, Blaszczyk R, Kaplon-Cieslicka A, Gawalko M, Tokarek T, Rajtar-Salwa R, Bil J, Wojewodzki M, Szpotowicz A, Krzciuk M, Bednarski J, Bakula-Ostalska E, Tomaszuk-Kazberuk A, Szyszkowska A, Welnicki M, Mamcarz A, Wozakowska-Kaplon B. Antithrombotic therapy in patients with atrial fibrillation undergoing percutaneous coronary intervention, including compliance with current guidelines-data from the POLish Atrial Fibrillation (POL-AF) Registry. Cardiovasc Diagn Ther. 2021 Feb;11(1):14-27. doi: 10.21037/cdt-20-839. PMID 33708474